CLINICAL TRIAL: NCT01799447
Title: The Relations Between Infants and Vulnerable First Time Mothers. Does Video Guidances With the Marte Meo Method Promote the Process? Intervention Study in a Community Setting
Brief Title: Early Intervention With the Marte Meo Method
Acronym: TiMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry); Region MidtJylland Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TiMM, AU, NN, FiM
Record Dates: First submitted 2013-02-06; First posted 2013-02-26 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Health Behavior; Mother-Child Relations
Keywords: Early intervention; Intervention study; Infant mother relations; First time mothers; Parental program; Marte Meo method; Video guidances
MeSH Terms: conditions — Health Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early intervention (Other): Early intervention. Quasiexperimental study. Inclusion of 150 first times families in intervention and matched with 150 families from control group.
  Interventions: Behavioral: Early intervention

INTERVENTIONS:
Behavioral: Early intervention — Interventions by health visitors with 18 months training in the Marte Meo method in order to promote relations between parents and infants.
  Other Names: Video gudiance with the Marte Meo method; Relations between infants and vulnerable first times mothers

SUMMARY:
Early intervention with the Marte Meo method. Aim to study whether the program have effect on:

Maternal confidence, maternal stress, maternal mood (EPDS), dyadic synchrony (Infant care index), and infants social competences (ASQ:SE)

DETAILED DESCRIPTION:
Relations between infant and vulnerable first time's mothers - Does video guidance with the Marte Meo method promote the process? Intervention study in a community setting

Background Infants develop their mentality, social and psychologically competencies in relations with parents and sensitive and responsive caregiving is important for infant's healthy development. Maternal responsiveness defined as the mother's ability to recognise infant's cues and act on those is a key to promote a secure child. At risk are unsecure/uncertain mothers, postpartum depressed mothers, mothers with preterm children and infants who in the perspective of the mother cries persistent and/or does not sleep well.

Danish public health nurses do home-visiting parents and they have opportunity to support parents in the development of relations to the infants. Some nurse's uses video-guidance with the Marte Meo method to promote the development of a healthy parent-infant relations, but knowledge about the effect of parent's having received video-guidance with the method is lacking.

Study part 1 Aim: To develop a screening tool to help public health nurses to identify unsecure mothers.

Design: Intervention Mapping step 1. Need assessment and development of few questions as a screening tool. Test of questions by face and content validation.

Study part 2 Develop a standardised preventive program step 2-4 in Intervention Mapping. The intervention is done by public health nurses, in home visits to first times mothers in the period from the child 2 to 6 months aged. The intervention includes 2-5 home visits with video-guidance's and has focus on the mother's ability to recognise infant's cues and act on those.

Excluded are families at sever risk who have been referred to treatment by psychiatric, psychological or social apartment.

Study 3 Test the program. Goal: to promote mothers parental self-efficacy, minimise mother's stress and mother's depressive mood. To promote infants social competences and promote mothers responsiveness and interaction with the infant.

Design: Quasi-experimental design. The intervention within 5 municipals with 36 "interventions public health nurses" (having a 1 ½ year educations as a Marte Meo therapist) and 85 "control public health nurses" who works as usually. The intervention group will includes 60 families and they will be matches with 60 families from the control groups.

Test: All first times mothers in the 5 municipals, when the children are 8 weeks old and after the intervention has stopped, when the children are 6 months old.

Test: All public health nurses when the interventions start and when the intervention stops.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers with children 7,8,9 weeks old.
* Mothers with EPDS from 8 to 13.
* Mothers who have delivered moderate to early between 32 and 37 weeks.
* And mothers with low maternal confidence

Exclusion Criteria:

* Mothers severe at risk, if they has been refereed to other departments than health nurses for treatment.

Ages: 7 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Child ASQ:SE | 3 month and 6 months
  Maternal self reported questionnaire when the child is 3 months old and when the child is 6 months old.

SECONDARY OUTCOMES:
Maternal stress (PSS) and confidence (KPCS) | 3 months after delivery and 6 months after delivery
  Validated PSS and KPCS

OTHER OUTCOMES:
Infant CARE-Index | 6 months after delivery
  Infant care index coding of videorecordings of mother and infant

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus university, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kristensen IH, Simonsen M, Trillingsgaard T, Kronborg H. Video feedback promotes relations between infants and vulnerable first-time mothers: a quasi-experimental study. BMC Pregnancy Childbirth. 2017 Nov 15;17(1):379. doi: 10.1186/s12884-017-1568-1. PMID 29141587